CLINICAL TRIAL: NCT05097196
Title: Effects of Home Based Step Aerobic Exercises on the Functional Capacity and Physical Performance of Sedentary Young Adults: A Pilot Study
Brief Title: Effects of Home Based Step Aerobic Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yunus Emre Kundakçı, Lecturer, PhD, Afyonkarahisar Health Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/439
Record Dates: First submitted 2021-09-26; First posted 2021-10-28 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-05

CONDITIONS: Aerobic Exercise
Keywords: home-based exercise; step-aerobic exercise; wearable technology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Step Aerobic Group (Experimental): Step aerobic exercise
  Interventions: Other: Moderate-intensity aerobic activities

INTERVENTIONS:
Other: Moderate-intensity aerobic activities — The exercise intensity of the individual is planned at 50-60% heart rate reserve using the Karvonen method.

SUMMARY:
The aim of this study is to determine the effects of commercially produced new generation smart step board and step-aerobic exercises for 6 weeks on the functional capacity and physical performance of young sedentary individuals.

DETAILED DESCRIPTION:
The aim of this study is to determine the effects of commercially produced new generation smart step board and step-aerobic exercises for 6 weeks on the functional capacity and physical performance of young sedentary individuals. The primary outcomes to be evaluated are the functional improvements in individuals' balance, functional capacity, muscle strength, and resting heart rate after 6 weeks of step-aerobic exercises. Secondary results are the evaluation of the effects of individuals on jumping performance and exercise motivation. It is thought that the results obtained in the study will reveal new information for studies investigating home-based exercise and rehabilitation practices and may provide evidence for larger studies involving a diagnosis of a disease in the future.

ELIGIBILITY:
Inclusion Criteria:

* Not participating in an exercise program that is followed regularly for at least 6 months
* Able to use a wearable device and willing to regularly step aerobic exercise
* In possession of a smart phone, tablet or computer
* BMI 25 to 40 kg/m2

Exclusion Criteria:

* Severe concomitant diseases: chronic heart failure, liver cirrhosis, kidney failure, active cancer, and cardiovascular, orthopedic, neurological psychological other diseases
* Not continuing the exercise program for more than three
* Loss of balance due to loss of consciousness or dizziness in the last 6 months

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Functional capacity | 10 weeks
  Six minute walk test (6MWT) distance of the participants will be evaluated using the G-Walk sensor system
Resting heart rate | 10 weeks
  Resting heart rate measurements are beats per minute taken in the morning

SECONDARY OUTCOMES:
Flamingo Balance Test | 10 weeks
  Static balances of the subjects will be determined with the Flamingo Balance Test.
Quadriceps Strength | 10 weeks
  Testing will be done at 90 degrees of knee flexion using Mechanical Push/Pull Dynamometer (MPPD) 22 lb (Fabrication Enterprises Inc., USA).
Counter movement jump | 10 weeks
  The jump parameters of the participants will be evaluated using the G-Walk sensor system (BTS G-Walk BTS Bioengineering Company, Italy).
Exercise motivation | 10 weeks
  Motivation will be measured after exercise using a visual analog scale consisting of a 100 mm line. Individuals will mark on the line how motivated they are during exercise. Motivation points will be obtained by measuring the distance from zero to point o

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Emre Kundakci, PhD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Turkey (Türkiye)